CLINICAL TRIAL: NCT00504543
Title: A 12 Month Open-label, Randomized, Multicenter, Sequential Cohort-group, Dose Finding Study to Evaluate the Efficacy, Safety and Tolerability of Oral AEB071 Versus Cyclosporine in Combination With Everolimus, Basiliximab and Corticosteroids in de Novo Adult Renal Transplant Recipients.
Brief Title: Efficacy, Safety and Tolerability of AEB071 Versus Cyclosporine in the Novo Renal Transplant Recipients
Acronym: AEB071
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAEB071A2206
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplant, AEB071
MeSH Terms: interventions — sotrastaurin; Everolimus; Cyclosporine

ARMS (3):
- Neoral (Active Comparator)
  Interventions: Drug: Neoral
- AEB071 high dose with Cetican reduced dose (Active Comparator)
  Interventions: Drug: AEB071; Drug: Certican
- AEB071 low dose with Cetican standard dose (Active Comparator)
  Interventions: Drug: AEB071; Drug: Certican

INTERVENTIONS:
Drug: AEB071 — oral, twice daily
  Arms: AEB071 high dose with Cetican reduced dose; AEB071 low dose with Cetican standard dose
Drug: Certican — twice daily
  Arms: AEB071 high dose with Cetican reduced dose; AEB071 low dose with Cetican standard dose
Drug: Neoral — twice daily
  Arms: Neoral

SUMMARY:
This study will assess safety and efficacy of AEB071 combined with everolimus in a CNI-free (calcineurin inhibitor) regimen in renal transplant recipients.

ELIGIBILITY:
Inclusion criteria

* Male and female patients 18 years or older
* Recipients of first kidney transplant from a deceased or living not related donor

Exclusion criteria

* Need for medication prohibited in the study
* Patients with heart disease (own or family history)
* Patients or donor HIV, Hepatitis B (HBsAg) or Hepatitis C (HCV) positive
* Patients with high immunological risks
* Patients with a history of cancer
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2007-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Primary efficacy failure, defined as a composite efficacy endpoint of treated biopsy proven acute rejection,(BPAR) graft loss, death or loss to follow-up, 3 months after transplantation. | 12 months

SECONDARY OUTCOMES:
Primary efficacy failure endpoint,defined as a composite efficacy endpoint of treated(BPAR),graft loss, death or loss to follow-up of additional treatment regimen at Month 6; renal function at Month 3, Month 6 and Month 12 post transplant using GFR; PK | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (24):
- Argentina (2):
  - Argentina, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia, Sydney, Australia
- Austria (2):
  - Austria, Innsbruck
  - Austria, Wein
- Belgium, Ghent, Belgium
- Brazil, São Paulo, Brazil
- Colombia (2):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
- Czech Republic, Prague, Czechia
- France (2):
  - France, Lille
  - France, Toulouse
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Heidelberg
- Italy, Milan, Italy
- Netherlands, Rotterdam, Netherlands
- Norway, Oslo, Norway
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Košice
- Spain (2):
  - Spain, Barcelona
  - Spain, Madrid
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Taipie, Taiwan

REFERENCES:
- [Result] Tedesco-Silva H, Kho MM, Hartmann A, Vitko S, Russ G, Rostaing L, Budde K, Campistol JM, Eris J, Krishnan I, Gopalakrishnan U, Klupp J. Sotrastaurin in calcineurin inhibitor-free regimen using everolimus in de novo kidney transplant recipients. Am J Transplant. 2013 Jul;13(7):1757-68. doi: 10.1111/ajt.12255. Epub 2013 May 9. PMID 23659755